CLINICAL TRIAL: NCT05482139
Title: Incisional Hernia Repair With Mesh at Waitemata District Health Board - A 15 Year Retrospective Cohort Study'
Status: Completed | Type: Observational
Sponsor: Waitemata District Health Board (Other Government)
Responsible Party: Principal Investigator, Alina Rankin, Non SET Surgical Registrar, Waitemata District Health Board
Other Study IDs: RM14763
Record Dates: First submitted 2022-07-16; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Incisional hernia repair with mesh — open or laparoscopic repairs of incisional hernia with mesh

SUMMARY:
A retrospective review of all incisional hernia repairs at North Shore Hospital (NSH), Auckland, NZ was performed between January 2004 and July 2019. Patients who had an open or laparoscopic incisional hernia repair with mesh were included in this study. Patients were retrospectively followed up from the date of their operation until the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Primary surgical procedure was incisional hernia repair with mesh

Exclusion Criteria:

* Suture repair
* Other hernia repair (not incisional)
* Operation notes unavailable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who had an incisional hernia repair with mesh at WDHB between January 2004 and July 2019
Sampling Method: Non-Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Post operative complications | 30-days post procedure
  Post operative complications as per Clavien-Dindo classification
Length of Hospital Stay | 0 days - 38 days
  How long patients stayed admitted to hospital after surgery

SECONDARY OUTCOMES:
Recurrence of hernia | 0 days - 15 years
  Did patients experience a recurrence of their hernia, if so after what period of time post operatively.

IPD SHARING:
Plan to Share IPD: No